CLINICAL TRIAL: NCT05879172
Title: Application of Electric Tubular Anastomotic Device in Colorectal Tumor Surgery: a Multi-center Clinical Trial
Brief Title: Electric Tubular Anastomosis in Rectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LI XIN-XIANG (Other)
Responsible Party: Sponsor-Investigator, LI XIN-XIANG, Professor, Fudan University
Organization: Fudan University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FDCRC71-LXX
Record Dates: First submitted 2023-05-07; First posted 2023-05-30 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Anastomosis; Rectal Cancer
Keywords: electric tubular anastomotic device
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- traditional anastomotic device (Active Comparator)
  Interventions: Device: traditional anastomotic device
- electric tubular anastomotic device (Experimental)
  Interventions: Device: electric tubular anastomotic device

INTERVENTIONS:
Device: electric tubular anastomotic device — The electric tubular anastomotic device developed by Suzhou Yingtukang Medical Technology Co., Ltd. is used for colorectal end-to-end and end-to-side anastomosis. This product is suitable for open or minimally invasive colorectal cancer surgery.
  Before firing the device, tissue thickness should be carefully assessed to prevent poor staling leading to leakage, inadequate hemostasis, or poor treatment.
  Arms: electric tubular anastomotic device
Device: traditional anastomotic device — Traditional anastomosis is used in this group. Staplers of the same brand are uniformly adopted to avoid differences between groups caused by different brands.
  Arms: traditional anastomotic device

SUMMARY:
Compared with traditional manual suturing, mechanical anastomosis can reduce the error caused by human factors. The electric anastomotic device can improve the automation and accuracy of anastomosis, reduce the requirements for doctors' operation, and establish a more standardized usage specification, thereby reducing the surgical complication rate and improving the quality of anastomosis. The clinical study of electric tubular anastomotic device adopts a multicenter, randomized, parallel controlled non-inferior study design, and randomly groups according to the 1:1 ratio to evaluate the clinical effectiveness and safety of electric tubular anastomotic device compared with conventional manual device.

DETAILED DESCRIPTION:
Compared with traditional manual suturing, mechanical anastomosis can reduce the error caused by human factors, involving the advantages like simple operation, short operation time, fast postoperative recovery, etc. Mechanical anastomosis can also ensure the consistency and repeatability of the surgical anastomosis process. The electric anastomotic device can improve the automation and accuracy of anastomosis, reduce the requirements for doctors' operation, and establish a more standardized usage specification, thereby reducing the surgical complication rate and improving the quality of anastomosis.

The clinical study of electric tubular anastomotic device adopts a multicenter, randomized, parallel controlled non-inferior study design, and randomly groups according to the 1:1 ratio to evaluate the clinical effectiveness and safety of electric tubular anastomotic device compared with conventional manual device.

The effectiveness of the electric tubular anastomotic device was evaluated by taking the success rate of anastomosis and anastomosis-related adverse events as the main evaluation indexes, while the operation performance evaluation, operation time, anastomosis time and postoperative recovery as the secondary evaluation indicators. The safety of electric tubular anastomotic device was evaluated by adverse events, vital signs, laboratory tests, etc.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-80y;
* Patients with resectable rectal cancer who are scheduled to undergo Dixon surgery (definition of rectal cancer: the lower boundary of the tumor is 10 cm from the anus≤);
* The patient consents to participate in the clinical study and signs the informed consent form.

Exclusion Criteria:

* Patients with significant local or systemic severe infection;
* Acute abdomen: intestinal obstruction, peritonitis, intestinal perforation;
* Have a systemic underlying disease that has not been controlled, or is unstable; Patients with poor constitution or serious other organic diseases who cannot tolerate anesthesia and surgery;
* Women during pregnancy, perinatal and lactation;
* Patients who are mentally incapable or unable to understand the requirements of the study;
* Patients who participated in other clinical studies 6 weeks before the start of this study or at the same time;
* The life expectancy of patients with malignant tumors is less than 6 months;
* Those who are critically ill and find it difficult to make an accurate evaluation of the effectiveness and safety of the device;
* Patients with diseases who are believed not suitable to participate in this clinical study;
* Have other diseases that are against anastomosis;
* The patient is receiving hormone therapy or immunosuppressive therapy;
* Albumin< 30g/dl.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
success rate of anastomosis | 1 week after surgery
  The end-to-end and end-to-side anastomosis of the intestinal tissue is performed during the operation. After the performance of anastomosis, the instrument is withdrawn. The anastomosis should be checked of accuracy, completeness and bleeding.

SECONDARY OUTCOMES:
time period of anastomosis | during the operation
time period of recovery | 1 year after surgey
  time of first postoperative defecation or exhausting

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China